CLINICAL TRIAL: NCT06946875
Title: The Effect of Pain Intensity, Neck Disability, Anxiety, and Quality of Life on Pain Threshold in Young Adults With Chronic Neck Pain
Brief Title: Factors Associated With Pain Threshold in Young Adults With Chronic Neck Pain
Status: Completed | Type: Observational
Sponsor: KTO Karatay University (Other)
Responsible Party: Sponsor
Other Study IDs: KaratayUBD1
Record Dates: First submitted 2025-04-21; First posted 2025-04-27 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-04

CONDITIONS: Neck Pain Chronic
MeSH Terms: interventions — Pain Threshold

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort1-Chronic Neck Pain Group: All participants have chronic neck pain and will be evaluated observationally.
  Interventions: Other: Pain Threshold

INTERVENTIONS:
Other: Pain Threshold — The pain thresholds of the participants will be measured with an algometer device. With this device, the minimum pressure threshold that causes pain is recorded.

SUMMARY:
The aim of this study was to determine which factors affect treatment expectations in individuals with chronic neck pain.

DETAILED DESCRIPTION:
This study aims to investigate the factors influencing treatment expectations in individuals suffering from chronic neck pain. Neck pain is a prevalent musculoskeletal disorder that significantly affects individuals' quality of life over long periods. It is recognized globally as the fourth leading cause of disability and imposes substantial economic burdens due to treatment costs, loss of workforce productivity, and healthcare expenditures.

Chronic neck pain often arises from nonspecific mechanical and postural causes, with various risk factors including socio-demographic (age, gender, genetics, obesity, occupation), psychological (stress, anxiety, depression, personality traits), and behavioral (postural disorders, prolonged sedentary work positions, smoking, physical activity habits) contributing to its development.

Pain duration classification categorizes neck pain as acute (up to six weeks), subacute (six weeks to three months), and chronic (over three months). The prevalence of chronic neck pain is increasing due to technological advancements and lifestyle changes, such as prolonged phone and computer use.

Psychological factors play a significant role in chronic neck pain, with high rates of depression and anxiety observed among affected individuals. These psychosocial factors, along with pain severity and disability, adversely impact patients' quality of life and pain threshold levels.

Despite extensive research, there is a lack of studies examining the combined effects of pain severity, neck disability, anxiety, and quality of life on pain threshold among young adults with chronic neck pain. This study seeks to fill this gap by exploring these relationships, aiming to contribute to the literature and support the development of a multidisciplinary approach to neck pain treatment.

ELIGIBILITY:
Inclusion Criteria:

* to be examined by specialised physicians and diagnosed with chronic neck pain
* to be physically and mentally fit to participate in the study.

Exclusion Criteria:

* the presence of instability in the neck joints,
* trauma within the last year,
* severe osteoporosis,
* previous neck surgery,
* physical therapy within the last 6 months,
* neurological findings or radiculopathy were determined.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Young Adults with Chronic Neck Pain
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Pain Threshold | Baseline
  The pain thresholds of the participants will be measured with an algometer device. With this device, the minimum pressure threshold that causes pain is recorded. Algometer is used as a standard in pain and sensorial threshold measurements (24). Pain threshold measurements will be performed on the specified point in all patients. Measurements will be made with a 1 cm² disc head apparatus connected to a pressure device calibrated to kg/cm² in power unit. The patient will be instructed to give the 'stop' command at the first sensation of pain. The applied pressure will be increased until the patient first feels the pain. The measurement will be terminated with the patient's stop command. Measurements were made 3 times from the same point and their average will be taken.
  The pressure pain threshold will be evaluated as the centre of the upper trapezius muscle.

SECONDARY OUTCOMES:
Visual Analogue Scale | Baseline
  The scale used in pain assessment, the Visual Analogue Scale, consists of a 10 cm horizontally positioned line on the page. The number '0', which is the starting point on this line, represents that the patient does not feel any pain, and the number '10' represents the worst pain experienced by the patient within their own experience. The patient is asked to mark any place he/she wants on this straight line between 0 and 10 in order to show the pain he/she has at the time the test is applied. Then, with the help of a ruler, the distance of the point marked by the patient to the starting point, the number 0, is measured and the value obtained is recorded.
Neck Disability Index | Baseline
  The Neck Disability Index (NDI) consists of 10 items: pain intensity, personal care, lifting, reading, headache, concentration, working, driving, sleeping and recreation. The individuals included in the study were asked to give a score between 0 (no disability) and 5 (full disability) for each item. For each answer option, A: 0 points, B: 1 point, C: 2 points, D: 3 points, E: 4 points, F: 5 points were calculated. The total score ranges from 0 (no disability) to 50 (full disability).
  * 0-4: no disability 22
  * 5-14: mild disability
  * 15-24: moderate disability
  * 25-34: severe disability
  * 35-50: considered as totally disabled.
Nottingham Health Profile | Baseline
  The Nottingham Health Profile is a 38-question general quality of life questionnaire developed to examine perceived health problems and the extent to which these problems affect activities of daily living. The questionnaire has a total of 6 sub-headings including 3 questions for energy level, 8 for pain, 9 for emotional reactions, 5 for sleep, 5 for social isolation and 8 for physical mobility. Each sub-heading is worth a total of 100 points and the value of each question is determined by dividing this value by the number of questions of the relevant section. A 'yes' answer to the questions is worth the score of the question, while a 'no' answer is worth zero points.
Beck Anxiety Scale | Baseline
  The questions in the Beck anxiety scale are related to anxiety symptoms. In the scale consisting of 21 questions in total, each question has four options in total as 'none, mild, moderate, severe'. The evaluation of the questions is done by considering the last week. Turkish adaptation, validity and reliability studies were conducted

CONTACTS AND LOCATIONS:
Overall Officials: Burcu DURSUN, Lecturer, Principal Investigator — KTO Karatay University
Locations (1):
- Kto Karatay Üniversitesi, Karatay, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No